CLINICAL TRIAL: NCT01631942
Title: A Multi-centre, Open Labelled, Multiple Dosing Trial Investigating Safety, Pharmacokinetics and Pharmacodynamics of NNC 0172-2021 Administered Subcutaneously to Healthy Male Subjects and Haemophilia Subjects
Acronym: explorer™2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7415-3986; 2011-005757-32 (EudraCT Number); U1111-1126-0327 (Other: WHO)
Record Dates: First submitted 2012-06-28; First posted 2012-06-29 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Healthy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose (healthy subjects) (Experimental)
  Interventions: Drug: NNC172-2021
- Medium dose (subjects with haemophilia) (Experimental)
  Interventions: Drug: NNC172-2021
- High dose (subjects with haemophilia) (Experimental)
  Interventions: Drug: NNC172-2021

INTERVENTIONS:
Drug: NNC172-2021 — Administered as subcutaneous (s.c., under the skin) injections every other day for two weeks.
  Escalation to next dose level is based on a safety evaluation.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate safety, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of NNC 0172-2021 administered subcutaneously to healthy male subjects and subjects with haemophilia.

DETAILED DESCRIPTION:
The present phase 1 trial has been terminated due to the need for changes in the trial design requiring a new re-designed multiple dosing phase 1 trial. Initiation of this new trial awaits additional non-clinical data.

ELIGIBILITY:
Inclusion Criteria:

* For haemophilia subjects only: Subjects diagnosed with haemophilia A with a baseline level of Factor VIII or Factor IX below 2% without inhibitors

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products
* Thrombocyte count below the lower limit of normal range at screening
* Any clinical signs or known history of thromboembolic events, or subject considered at high risk of thromboembolic events as judged by the investigator or subjects at increased risk of cardiovascular disease as judged by the investigator

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2012-06-26 (Actual); Primary Completion 2012-09-04 (Actual); Study Completion 2012-09-04 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | From first trial drug administration through trial day 35

SECONDARY OUTCOMES:
Local tolerability | After the last s.c. dose administration (trial day 15)
Thrombocyte count | After the last s.c. dose administration (trial day 15)
Trough level (Ctrough) | Prior to the last s.c. dose administration (trial day 15)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (6):
- Novo Nordisk Investigational Site, Vienna, Austria
- France (2):
  - Novo Nordisk Investigational Site, Lyon
  - Novo Nordisk Investigational Site, Montpellier
- Novo Nordisk Investigational Site, Berlin, Germany
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Harrow, United Kingdom

REFERENCES:
- [Result] Waters EK, Sigh J et al.: Trombin generation is increased in plasma from healthy males who have received concizumab, an antibody against tissue factor pathway inhibitor (ExplorerTM 2); Journal of Thrombosis and Haemostasis, Abstracts 2015; 13(Suppl. S2): 1-997(AS019)
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com